CLINICAL TRIAL: NCT07249671
Title: Effects of Rope Skipping in Cardiopulmonary Fitness in School Going Children
Brief Title: Effects of Rope Skipping in Cardiopulmonary Fitness in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: : REC/RCR&AHS/MOIZAKHAN
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cardiopulmonary
Keywords: Cardiopulmonary, rope skipping, Borg scale.

STUDY DESIGN:
Intervention Model Description: The study will be conducted in a school setting, involving a randomized control trial (RCT) of 178 children aged 6 to 12. The participants will be divided into two groups: a control group engaging in regular physical education (PE) classes and an experimental group practicing rope skipping for 50 minutes, three times a week, over a period of 8 weeks. Cardiopulmonary fitness will be assessed before and after the intervention using the borg rating scale and talk test of perceived exertion.. Data will be analyzed to determine changes in endurance, heart rate recovery, and lung function between the groups. The expected outcome is a significant improvement in cardiopulmonary parameters among the rope-skipping group, highlighting the exercise's effectiveness in promoting heart and lung health in children.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Intervention Group ( Rope Skipping) (Active Comparator): rope skipping exercise performed 50 minutes/time (including warmup and cool down session) 3 times/ week for 8 weeks
  Interventions: Other: Rope skipping
- Group B : Control Group ( Self directed unsupervised free play) (Active Comparator): The control group was engaged in self directed unsupervised free play for 50 minutes/time.
  3 times/ week for 8 weeks
  Interventions: Other: unsupervised free play

INTERVENTIONS:
Other: Rope skipping — Rope skipping exercise performed 50 minutes/ times ( including warm up and cool down session) 3 times / week for 8 weeks
  Arms: Group A: Intervention Group ( Rope Skipping)
Other: unsupervised free play — The control group was engaged in self directed unsupervised free play.
  Arms: Group B : Control Group ( Self directed unsupervised free play)

SUMMARY:
The study will be conducted in a school setting, involving a randomized control trial (RCT) of 178 children aged 6 to 12. The participants will be divided into two groups: a control group engaging in regular physical education (PE) classes and an experimental group practicing rope skipping for 50 minutes, three times a week, over a period of 8 weeks. Cardiopulmonary fitness will be assessed before and after the intervention using the borg rating scale and talk test of perceived exertion.. Data will be analyzed to determine changes in endurance, heart rate recovery, and lung function between the groups. The expected outcome is a significant improvement in cardiopulmonary parameters among the rope-skipping group, highlighting the exercise's effectiveness in promoting heart and lung health in children.

DETAILED DESCRIPTION:
Physical inactivity among school-going children is a growing concern globally, leading to increased risks of cardiovascular diseases, obesity, and poor overall health. Cardiopulmonary fitness, an important indicator of a healthy heart and lungs, can significantly reduce these risks. Rope skipping, a simple yet effective exercise, is gaining attention as a potential intervention to enhance cardiopulmonary fitness in children. Its low cost, accessibility, and high intensity make it a feasible activity in school environments. This project investigates the impact of regular rope skipping on the cardiopulmonary fitness of school-going children, aiming to assess improvements in heart rate, endurance, and respiratory capacity. By evaluating these parameters, the study seeks to contribute to the growing body of evidence supporting physical activity as a crucial part of children's health routines.

The study will be conducted in a school setting, involving a randomized control trial (RCT) of 178 children aged 6 to 12. The participants will be divided into two groups: a control group engaging in regular physical education (PE) classes and an experimental group practicing rope skipping for 50 minutes, three times a week, over a period of 8 weeks. Cardiopulmonary fitness will be assessed before and after the intervention using the borg rating scale and talk test of perceived exertion.. Data will be analyzed to determine changes in endurance, heart rate recovery, and lung function between the groups. The expected outcome is a significant improvement in cardiopulmonary parameters among the rope-skipping group, highlighting the exercise's effectiveness in promoting heart and lung health in children.

ELIGIBILITY:
Inclusion Criteria:

* School going children age 6 to 12 years
* Children with no pre existing regular rope skipping training
* No student athletes
* Children with no physical and psychological disabilities

Exclusion Criteria:

* Children with pre existing injuries
* Children with chronic medical conditions
* Children with cardiovascular issues
* Children with disability

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 178 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Borg rating scale | duration 8 weeks
  The original Borg scale ranges from 6 to 20, where 6 represents "no exertion at all" and 20 represents "maximal exertion.
Talk test of Perceived Exertion | duration 8 weeks
  The Talk Test is a simple way to measure exercise intensity based on how easily a person can talk during activity
20 Meter Shuttle Run Test. | duration 8 weeks
  The 20 meter shuttle run test also know as beep test is a field test that measures aerobic fitness and predicts the maximal rate of oxygen consumption (VO2max)

CONTACTS AND LOCATIONS:
Overall Officials: Moiza Khan, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Allied school, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powell TA, Mysliwiec V, Brock MS, Morris MJ. OSA and cardiorespiratory fitness: a review. J Clin Sleep Med. 2022 Jan 1;18(1):279-288. doi: 10.5664/jcsm.9628. PMID 34437054